CLINICAL TRIAL: NCT02633631
Title: The Center for Contraceptive Excellence: an Innovative Health Services Delivery and Payment Model
Brief Title: Contraceptive Choice Center
Acronym: C3
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Centers for Medicare and Medicaid Services (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 201410028
Record Dates: First submitted 2015-04-22; First posted 2015-12-17 (Estimated); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Unintended Pregnancy; Contraception; Family Planning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women seeking family planning services: Women seeking family planning and gynecological services will be enrolled in our study.

SUMMARY:
The Contraceptive Choice Center will use an innovative-model of contraceptive care which was developed as a part of the Contraceptive CHOICE Project (CHOICE). This delivery model will deliver high-quality family planning services for women and reduce unintended pregnancies and births. This intervention will result in improved health for women, improved health care, and reduced costs to Medicaid.

The Center will provide care to women ages 14-45 years of age.

DETAILED DESCRIPTION:
The Center will provide high-quality contraceptive care using the innovative model of the Contraceptive CHOICE Project. Specifically, the model will provide the following components: 1) Structured, evidence-based contraceptive counseling; 2) education of providers about long-acting reversible contraceptive (LARC) methods and evidence-based guidelines for contraceptive provision; 3) removal of patient barriers to family planning services; and 4) post-visit contraceptive support. The model addresses the barriers to contraceptive uptake.

ELIGIBILITY:
Inclusion Criteria:

* Childbearing-age seeking family planning services
* Negative pregnancy test
* Willing and able to undergo informed consent

Exclusion Criteria:

* Current participation in a research study that would interfere with the conduct of this study
* Currently pregnant

Ages: 14 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: We plan to recruit women who are at high risk for unintended pregnancy and birth.
Sampling Method: Non-Probability Sample
Enrollment: 2664 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Rate of unintended pregnancy | 24 months
  Reduce unintended pregnancy by 10% - # of pregnancies that are unintended per 1000 reproductive-age women (14-45 years)

SECONDARY OUTCOMES:
Rate of unintended births | 24 months
  Reduce unintended births and associated costs by 15% - # of births that are unintended per 1000 reproductive age women

CONTACTS AND LOCATIONS:
Overall Officials: Tessa Madden, MD,MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Division of Clinical Research at Washington University, St Louis, Missouri, United States